CLINICAL TRIAL: NCT02536794
Title: A Single Arm Phase II Study Evaluating the Efficacy and Safety of MEDI4736 in Combination With Tremelimumab in Patients With Metastatic Her2 Negative Breast Cancer
Brief Title: MEDI4736 and Tremelimumab in Treating Patients With Metastatic HER2 Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: MedImmune LLC (Industry); Avon Breast Cancer Foundation (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 15B01; NCI-2015-01445 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ESR-14-10694; D4190C00030; STU00200984; NU 15B01 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Results first posted 2021-04-23 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-04

CONDITIONS: Estrogen Receptor Negative; Estrogen Receptor Positive; HER2/Neu Negative; Recurrent Breast Carcinoma; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (MEDI4736, tremelimumab) (Experimental): Patients receive anti-B7H1 monoclonal antibody MEDI4736 IV over 1 hour and tremelimumab IV over 1 hour on day 1. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Four weeks after the last combination dose, patients continue to receive anti-B7H1 monoclonal antibody MEDI4736 every 2 weeks for up to 18 additional doses in the absence of disease progression or unacceptable toxicity. Patients achieving PD or clinical benefit (CR, PR, or SD) may be retreated with anti-B7H1 monoclonal antibody MEDI4736 for an additional 52 weeks.
  Interventions: Biological: Anti-B7H1 Monoclonal Antibody MEDI4736; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Biological: Tremelimumab

INTERVENTIONS:
Biological: Anti-B7H1 Monoclonal Antibody MEDI4736 — Given IV
  Other Names: MEDI4736
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP-675; CP-675,206; CP-675206; Ticilimumab

SUMMARY:
The main purpose of this study is to determine the anti-tumor activity of MEDI4736 in combination with tremelimumab in patients with metastatic HER2-negative breast cancer. Both MEDI4736 and tremelimumab are antibodies (proteins used by the immune system to fight infections and cancers). MEDI4736 attaches to a protein in tumors called PD-L1. It may prevent cancer growth by helping certain blood cells of the immune system get rid of the tumor. Tremelimumab stimulates (wakes up) the immune system to attack the tumor by inhibiting a protein molecule called CTLA-4 on immune cells. Combining the actions of these drugs may result in better treatment options for patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate clinical benefit rate in patients with metastatic HER2 negative breast cancer treated with MEDI4736 in combination with tremelimumab.

SECONDARY OBJECTIVES:

I. To evaluate progression free survival (PFS) and overall survival (OS) in patients with metastatic HER2 negative breast cancer treated with MEDI4736 in combination with tremelimumab.

II. To evaluate safety and tolerability.

TERTIARY OBJECTIVES:

I. To evaluate if tissue-based immunohistochemical expression of programmed death-ligand (PD-L)1; tumor infiltrating lymphocytes (TILs); peripheral T cell subpopulations; changes in tissue and peripheral T cell receptor genotype; human leukocyte antigen (HLA) genotype; and immune-related candidate gene signatures predict response to MEDI4736 in combination with tremelimumab.

II. To demonstrate the pharmacodynamic effects of MEDI4736 and tremelimumab on tissue and serum based biomarkers including PD-L1, TILs, T cell subpopulations, and T cell receptor genotype.

OUTLINE:

Patients receive MEDI4736 intravenously (IV) over 1 hour and tremelimumab IV over 1 hour on day 1. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Four weeks after the last combination dose, patients continue to receive MEDI4736 every 2 weeks for up to 18 additional doses in the absence of disease progression or unacceptable toxicity. Patients who achieve clinical benefit (complete response [CR], partial response [PR], or stable disease [SD]) until the end of the 52 week period will then enter follow-up. During follow-up patients who develop PD may be re-treated with MEDI4736 at the dose previously administered IV for an additional 52 weeks using the same guidelines as with the initial 52 week period if they meet treatment in the setting of PD criteria. Only one 52 week retreatment period will be allowed.

After completion of study treatment, patients are followed up at 3, 6, 9, and 12 months, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically documented (either primary or metastatic site) diagnosis of breast cancer that is HER2 non-overexpressing by immunohistochemistry, namely 0 or 1; if they have an equivocal immunohistochemistry, 2, the tumor must be non-gene amplified by fluorescence in situ hybridization (FISH) performed upon the primary tumor or metastatic lesion (ratio < 2 and HER2 copy number < 4); estrogen receptor (ER) positivity is defined as 1% or greater
* Patients must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Patients who are ER negative must have progressed through at least one prior chemotherapy regimen in the metastatic setting or within 12 months of their last adjuvant systemic treatment; patients who are ER positive must have progressed through standard hormone therapy options and have received at least one line of chemotherapy in the metastatic setting
* Completion of prior chemotherapy systemic anticancer therapy at least 2 weeks prior to study entry
* Radiation therapy must be completed at least 2 weeks prior to study entry; radiated lesions may not serve as measurable disease unless they have been radiated over 12 months prior to enrollment
* Patients may have parenchymal brain metastases if stable (no evidence of progression) for at least 1 month after local therapy (radiation or surgery); leptomeningeal disease is excluded; must have completed any prescribed steroid taper
* Patients may have had a prior diagnosis of cancer if it has been > 5 years since their last treatment
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 50,000/mcl
* Total bilirubin =< 1.5 times the institutional upper limit of normal (ULN) (or =< 3 times ULN in case of liver metastasis)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SPGT]) =< 2.5 X institutional ULN (or =< 5 times ULN in case of liver metastasis)
* Creatinine =< 2 ng/ml
* Females of child-bearing potential (FOCBP) and males must agree to use 2 methods of adequate contraception prior to study entry, for the duration of study participation, and for number (#) days following completion of therapy; should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

  * NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
  * Has not undergone a hysterectomy or bilateral oophorectomy
  * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* FOCBP must have a negative pregnancy test within 7 days prior to registration on study
* Willingness to provide a fresh biopsy prior to study enrollment and after 2 cycles of treatment
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier are not eligible.
* Current or prior use of immunosuppressive therapy within 2 weeks of starting investigational therapy
* Patients who are taking any herbal (alternative) medicines are NOT eligible for participation; patients must be off any such medications by the time of registration for at least 2 weeks; NOTE: Vitamin supplements are acceptable
* Patients may not have received any other investigational agents within 4 weeks prior to registration
* Prior treatment with immune therapy (including but not limited to cluster of differentiation [CD]137, OX40, programmed death [PD]-1, PD-L1 or cytotoxic T-lymphocyte antigen 4 [CTLA4] inhibitors)
* Prior severe infusion reaction to a monoclonal antibody
* Patients with a history of or active autoimmune disease within the past 3 years with the following exceptions:

  * Vitiligo or alopecia
  * Hypothyroidism on stable doses of thyroid replacement therapy
  * Psoriasis not requiring systemic therapy within the past 3 years
* History of primary immunodeficiency disease or tuberculosis
* Major medical conditions that might affect study participation (uncontrolled pulmonary, renal, or hepatic dysfunction, uncontrolled infection) are not eligible; other significant comorbid condition which the investigator feels might compromise effective and safe participation in the study
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Uncontrolled pulmonary, renal, or hepatic dysfunction
  * Ongoing or active infection requiring systemic treatment
  * Known active or chronic viral hepatitis or human immunodeficiency virus (HIV)
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Female patients who are pregnant or nursing are not eligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2021-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Santa-Maria, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Northwestern University- Lake Forest Hospital, Lake Forest, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was opened to accrual on December 18 2015, with the first patient starting treatment on January 14, 2016 and a total accrual goal of 50 patients. The study closed to further accrual July 20, 2020 with 30 patients treated on study.
Period: Reached 1st Response Assessment
Arm/Group | Treatment (MEDI4736, Tremelimumab)
Started | 30
Started Treatment | 30
Attempted First Cycle | 30
Attempted Second Cycle | 24
Reached First Response | 24
Completed | 24
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Progressive Disease | 2
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1
Period: Continued Treatment After 1st Response
Arm/Group | Treatment (MEDI4736, Tremelimumab)
Started | 24
Went on to Start Cycle 3 | 16
Completed | 16
Not Completed | 8
Not completed — Progressive disease | 7
Not completed — Adverse Event | 1
Period: Follow up for 3 Years or Death
Arm/Group | Treatment (MEDI4736, Tremelimumab)
Started (All patients who are treated on study go into the follow up phase) | 29 (one patient did not go into follow up as treatment was discontinued due to a protocol violation)
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (MEDI4736, Tremelimumab)
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 53.0 [35 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 24
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
Received prior systemic therapies for breast cancer [Count of Participants; unit: Participants] | 30
Received prior chemotherapy [Count of Participants; unit: Participants]
  No | 1
  yes | 29
ER Status [Count of Participants; unit: Participants] — Estrogen Receptors (ER) status is determined the presence or absence of estrogen receptors in the breast cancer cells. ER positive is defined as 1% or greater.
  Participants
    Negative | 15
    Positive | 15
PR Status [Count of Participants; unit: Participants] — progesterone receptor (PR) status is determined by the presence or absence of progresterone receptors in the breast cancer cells. PR positive will be defined as a result of greater than 10%.
  Participants
    Negative | 22
    Positive | 8
Triple Negative Breast Cancer (TNBC) [Count of Participants; unit: Participants] — TBNC is breast cancer which is ER negative, PR negative and HER2 negative
  Participants
    No | 15
    Yes | 15
HER 2 Status [Count of Participants; unit: Participants] — Human epidermal growth factor receptor 2 (HER2) status is determined to be positive (if the protein HER2 is present) or negative (protein HER2 is not present/present in very low levels).
  Participants
    Positive | 0
    Negative | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) in Patients With Metastatic HER2 Negative Breast Cancer Treated With Durvalumab in Combination With Tremelimumab
Description: Overall response rate is defined as the number of patients with partial response (PR), plus those with complete response (CR) using the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 with the following definitions:
  Complete Response - Disappearance of all lesions Partial Response - At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to a maximum of 49 cycles where 1 cycle = 4 weeks for the first 4 cycles and than 1 cycle =2 weeks for 45 cycles
Population: number of HER2 negative breast cancer patients that met criteria to be evaluable for this endpoint
Measure: Number; unit: participants
Arm/Group | Treatment (MEDI4736, Tremelimumab)
Number analyzed (Participants) | 27
participants | 4

2. Primary Outcome: Overall Response Rate (ORR) in Patients With Triple Negative Breast Cancer (TNBC) Treated With Durvalumab in Combination With Tremelimumab
Description: Overall response rate is defined as the number of patients with partial response (PR), plus those with complete response (CR) using the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 with the following definitions:
  Complete Response - Disappearance of all lesions Partial Response - At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  TNBC = patients whose status for ER, PR and HER2 is negative
Time Frame: Up to a maximum of 49 cycles where 1 cycle = 4 weeks for the first 4 cycles and then 1 cycle = 2 weeks for up to 45 cycles
Population: number of triple negative breast cancer patients that met criteria to be evaluable for this endpoint
Measure: Number; unit: participants
Arm/Group | Treatment (MEDI4736, Tremelimumab)
Number analyzed (Participants) | 14
participants | 4

3. Secondary Outcome: Toxicity in Patients With Metastatic HER2 Negative Breast Cancer Treated With Durvalumab in Combination With Tremelimumab
Description: Toxicity will be evaluated by the number, frequency, and severity of adverse events as defined by the NCI Common Terminology Criteria for Adverse Events or CTCAE version 4.03
  Events that were considered to at least be possibly related to either study drugs are reported here and in general grading is as follows:
  Mild (grade 1): the event causes discomfort without disruption of normal daily activities Moderate (grade 2): the event causes discomfort that affects normal daily activities Severe (grade 3): the event makes the patient unable to perform normal daily activities or significantly affects his/her clinical status Life-threatening (grade 4): the patient was at risk of death at the time of the event Fatal (grade 5): the event caused death
Time Frame: Up to a maximum of 49 cycles where 1 cycle = 4 weeks for the first 4 cycles and than 1 cycle =2 weeks for 45 cycles
Measure: Number; unit: participants
Arm/Group | Treatment (MEDI4736, Tremelimumab)
Number analyzed (Participants) | 30
participants
  Grade 1 or 2 Adverse Event | 27
  Grade 3 or 4 Adverse Event | 12
  Grade 1 or 2 Serious Adverse Event | 6
  Grade 3 or 4 Serious Adverse Event | 7

4. Secondary Outcome: Overall Survival (OS) in Patients With Metastatic HER2 Negative Breast Cancer Treated With Durvalumab in Combination With Tremelimumab
Description: OS is defined as the time from treatment initiation until death due to any cause
Time Frame: Time from treatment initiation until 3 years post treatment continuation where patients were treated up to a maximum of 49 cycles where 1 cycle = 4 weeks for the first 4 cycles and than 1 cycle =2 weeks for 45 cycles
Population: number of HER2 negative breast cancer patients that met criteria to be evaluable for this endpoint
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (MEDI4736, Tremelimumab)
Number analyzed (Participants) | 27
months | 11.3 [7.16 to 36.6]

5. Secondary Outcome: Progression Free Survival (PFS) in Patients With Metastatic HER2 Negative Breast Cancer Treated With Durvalumab in Combination With Tremelimumab
Description: PFS is defined as the time from treatment initiation to documented disease progression. Progressive Disease is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression.)
Time Frame: Time from treatment initiation until 3 years post treatment continuation where patients were treated up to a maximum of 49 cycles where 1 cycle = 4 weeks,for the first 4 cycles and than 1 cycle =2 weeks for 45 cycles
Population: number HER2 negative breast cancer patients that met criteria to be evaluable for this endpoint
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (MEDI4736, Tremelimumab)
Number analyzed (Participants) | 27
months | 4.86 [3.09 to 7.89]

6. Secondary Outcome: Clinical Benefit Rate (CBR) in Patients With Metastatic HER2 Negative Breast Cancer Treated With Durvalumab in Combination With Tremelimumab
Description: CBR is defined as the number of patients with complete response (CR) plus those with partial response (PR) plus those with stable disease (SD) for ≥ 12 weeks using Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 with the following definitions:
  Complete Response - Disappearance of all lesions Partial Response - At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters Stable Disease - Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum of diameters while on study
Time Frame: Up to a maximum of 49 cycles where 1 cycle = 4 weeks for the first 4 cycles and than 1 cycle =2 weeks for 45 cycles
Population: Per protocol patients were required to complete 2 months of study treatment to be evaluable for this endpoint, however all patients who had a response are reported here as the study did not meet its total sample size. number of patients HER2 negative breast cancer patients that met criteria to be evaluable for this endpoint
Measure: Number; unit: participants
Arm/Group | Treatment (MEDI4736, Tremelimumab)
Number analyzed (Participants) | 27
participants | 5

7. Other Pre Specified Outcome: Tumor Infiltrating Lymphocytes (TILs) Expression
Description: To evaluate if tissue-based immunohistochemical expression of TILs predicts response to MEDI4736 in combination with tremelimumab. Changes will also be analyzed to assess for pharmacodynamic effects of treatment
Time Frame: Baseline and at 2 months of treatment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Programmed Death-ligand 1 (PD-L1) Expression
Description: To evaluate if tissue-based immunohistochemical expression of PD-L1 predicts response to MEDI4736 in combination with tremelimumab. Changes will also be analyzed to assess for pharmacodynamic effects of treatment
Time Frame: Baseline and at 2 months of treatment
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in T Cell Receptor Genotype
Description: To evaluate if tissue-based immunohistochemical expression of T cell receptor genotype predicts response to MEDI4736 in combination with tremelimumab. Changes will also be analyzed to assess for pharmacodynamic effects of treatment
Time Frame: Baseline and at 2 months of treatment
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Changes in Peripheral T Cell Subpopulations
Description: To evaluate if tissue-based immunohistochemical expression of peripheral T cell subpopulations predicts response to MEDI4736 in combination with tremelimumab. Changes will also be analyzed to assess for pharmacodynamic effects of treatment
Time Frame: Baseline and at 2 months of treatment
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Human Leukocyte Antigen (HLA)
Description: To evaluate if tissue-based immunohistochemical expression of HLA predicts response to MEDI4736 in combination with tremelimumab
Time Frame: Baseline and at 2 months of treatment
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Immune-related Candidate Gene Signatures
Description: To evaluate if tissue-based immunohistochemical expression of Immune-related candidate gene signatures predicts response to MEDI4736 in combination with tremelimumab
Time Frame: Baseline and at 2 months of treatment
Reporting Status: Not Posted

13. Post Hoc Outcome: Response in Patients With Metastatic HER2 Negative Breast Cancer Treated With Durvalumab in Combination With Tremelimumab
Description: Patients response is defined as the best response to treatment whilst on study using Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 with the following definitions:
  Complete Response - Disappearance of all lesions Partial Response - At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters Stable Disease - Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum of diameters while on study Progressive Disease - At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression.)
Time Frame: Up to a maximum of 49 cycles where 1 cycle = 4 weeks for the first 4 cycles and than 1 cycle =2 weeks for 45 cycles
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (MEDI4736, Tremelimumab)
Number analyzed (Participants) | 30
Participants
  Complete Response | 1
  Partial Response | 3
  Stable Disease | 4
  Progressive Disease | 19
  Not evaluable | 3

14. Post Hoc Outcome: Overall Response Rate (ORR) in Patients With Metastatic HER2 Negative Breast Cancer Treated With Durvalumab in Combination With Tremelimumab (All Included)
Description: as for outcome 1
Time Frame: Up to a maximum of 49 cycles where 1 cycle = 4 weeks for the first 4 cycles and than 1 cycle =2 weeks for 45 cycles
Population: This includes patients who did not complete 2 months of treatment but would otherwise be evaluable for the endpoint
Measure: Number; unit: participants
Arm/Group | Treatment (MEDI4736, Tremelimumab)
Number analyzed (Participants) | 27
participants | 4

ADVERSE EVENTS:
Time Frame: Adverse events are collected from the time of treatment initiation until 30 days post last treatment. Adverse events were collected up to a maximum of 49 cycles where 1 cycle = 4 weeks for the first 4 cycles and than 1 cycle =2 weeks for 45 cycles.
Arm/Group | Treatment (MEDI4736, Tremelimumab)
All-Cause Mortality (participants affected / at risk) | 22/30
Serious Adverse Events (participants affected / at risk) | 18/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (MEDI4736, Tremelimumab) (N=30)
Confusion (Nervous system disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 2 (2)
Myocarditis and Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Spontaneous bacterial peritonitis (Infections and infestations) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) — Patient also experienced diarrhea during this event
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 1 (1) — Patient also experienced pain during this event
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Patient also experienced hypersomnia during this event
Dizziness (Nervous system disorders) | 1 (1) — Patient also experienced headaches and vomiting at the time of this event
Fever and chills (General disorders) | 2 (2) — one patient also experienced elevated AST and hepatic hemorrhage at the time of the event
Fever (General disorders) | 1 (1) — Patient also experienced weakness at the time of the event
Enteritis (Gastrointestinal disorders) | 1 (1) — Patient also experienced increased INR at the time of the event
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Patient also experience anorexia and edema in limbs at the time of this event
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) — patient experienced pleural effusion and pneumonitis during this event
Pseudoprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Patient also experienced fever, left arm weakness and gait disturbance during this event
Urosepsis (Infections and infestations) | 1 (1) — Patient also experienced pain and delirium during this event
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (MEDI4736, Tremelimumab) (N=30)
Anemia (Blood and lymphatic system disorders) | 15
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 3
Ear pain (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 4
Blurred vision (Eye disorders) | 1
Floaters (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 8
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Colitis (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 6
Dry mouth (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Oral pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Chills (General disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 11
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 1
Night sweats (General disorders) | 1
Breast leison discomfort (General disorders) | 1
Discomfort (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 4
Pharyngitis (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 2
Vaginal infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 9
Alanine aminotransferase increased (Investigations) | 9
Alkaline phosphatase increased (Investigations) | 11
Aspartate aminotransferase increased (Investigations) | 9
Blood bilirubin increased (Investigations) | 7
Cardiac troponin I increased (Investigations) | 1
Creatinine increased (Investigations) | 3
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
GGT increased (Investigations) | 8
Hemoglobin increased (Investigations) | 1
INR increased (Investigations) | 4
low GFR (clinically significant) (Investigations) | 1
LV diastolic dysfunction (Investigations) | 1
Lipase increased (Investigations) | 6
Lymphocyte count decreased (Investigations) | 13
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 7
Serum amylase increased (Investigations) | 3
Weight gain (Investigations) | 1
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 2
Alkalosis (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 18
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 4
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 16
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 10
Hyponatremia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1
joint stiffness (feet) (Musculoskeletal and connective tissue disorders) | 1
generalized aches and pains (Musculoskeletal and connective tissue disorders) | 1
cancer related pain (Musculoskeletal and connective tissue disorders) | 1
bilateral hand stiffness (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Nervous system disorder NOS (Nervous system disorders) | 1
Ptosis (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Proteinuria (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Lymphedema (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
The study was closed before reaching the planned total sample size of 50 patients due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT02536794/Prot_SAP_000.pdf